CLINICAL TRIAL: NCT03518658
Title: BlueSync Field Evaluation
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: BlueSync Field Evaluation
Record Dates: First submitted 2018-04-20; First posted 2018-05-08 (Actual); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Bradycardia
Keywords: remote monitoring; transmission compliance; patient engagement
MeSH Terms: conditions — Bradycardia; Patient Participation | interventions — Control Groups; Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Evaluation Group: Patients implanted with a pacemaker or CRT-P device who will be using remote monitoring via the MyCareLink Heart App
  Interventions: Other: Evaluation Group
- Control Group: Patients with low power implantable devices and CareLink Monitor 2490 (Excluding wireless model 2490C)
  Interventions: Other: Control Group (Historical)

INTERVENTIONS:
Other: Evaluation Group — Patient receiving exposure to the MyCareLink Heart App during device pairing
  Groups: Evaluation Group
Other: Control Group (Historical) — Patients receiving exposure to the CareLink Monitor 2490 (Excluding wireless model 2490C). The patients' data will be extracted from Medtronic de-identified CareLink™ database.
  Groups: Control Group

SUMMARY:
The purpose of this field evaluation is to collect and evaluate information related to CareLink transmission compliance as well as patient perceived benefit of BlueSync™ and the health care provider perception of the value of BlueSync™ and satisfaction with BlueSync™.

DETAILED DESCRIPTION:
The primary goal is to learn how many CareLink quarterly scheduled transmissions are completed within a prescribed time period to assess CareLink scheduled transmission compliance. The evaluation will also assess adoption to remote monitoring, patient perceived benefit of BlueSync™ (how patients interact with the smart device application) and health care provider perception of the value of BlueSync™ and satisfaction with BlueSync™ (benefits experienced by clinicians that use BlueSync™).

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CRF 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CRF 11.24 and 11.44).

ELIGIBILITY:
Inclusion Criteria:

* Patient will be/has been implanted with an Azure™ or Percepta™, Serena™, Solara™ CRT-P device compatible with BlueSync™ (both new and replacement devices are allowed)
* Patient must own a smart device (Smartphone or tablet) that meets system requirements and be willing to use during evaluation period
* Patient must be able to complete the required 12-month follow-up after enrollment
* Patients must be of legal age according to local law

Exclusion Criteria:

* Patient unwilling to complete required surveys during 12-month evaluation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at hospitals and clinics specializing in the implant and followup of pacemakers and CRT-P devices using remote monitoring
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2019-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Trajki, MD, Principal Investigator — The Cleveland Clinic
Locations (20):
- United States (11):
  - Stanford Universithy, Palo Alto, California
  - Hartford Hosital, Hartford, Connecticut
  - Daytona Heart Group, Daytona Beach, Florida
  - Cardiovascular Institutes of Orland0, Orlando, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - CentraCare, Saint Cloud, Minnesota
  - The Valley Hospital, Ridgewood, New Jersey
  - Cone Health, Greensboro, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Mount Carmel, Columbus, Ohio
  - East Tennessee Consultants, Knoxville, Tennessee
- France (2):
  - CHU Bordeaux, Bordeaux
  - CHI Toulouse, Toulouse
- Italy (3):
  - Istituto clinico Città Studi, Milan
  - Ospedale Sacro Cuore, Negrar
  - Provincia Religiosa San Pietro Di Roma, Rome
- United Kingdom (4):
  - Sandwell and West Birmingham Hospitals, Birmingham
  - Manchester Royal Infirmary, Manchester
  - Southampton, Southampton
  - University Hospital of North Midlands NHS Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No
There are not plans to share IPD with other researchers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Historical Controls were not considered enrolled in this study. The patients' data was extracted from Medtronic de-identified CareLink™ database.
Groups:
- Control Group (Historical): Patients with low power implantable devices and CareLink Monitor 2490 (Excluding wireless model 2490C)
Period: Overall Study
Arm/Group | Evaluation Group | Control Group (Historical)
Started | 257 (Number of patients completing device pairing survey) | 128607
Completed | 206 (Number of patients completing annual survey) | 128607
Not Completed | 51 | 0
Not completed — Other | 51 | 0

BASELINE CHARACTERISTICS:
Population: Patients enrolled in the BlueSync Field Evaluation
Groups:
- Total: Total of all reporting groups
Arm/Group | Evaluation Group | Control Group (Historical) | Total
Number analyzed (Participants) | 257 | 128607 | 128864
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 50 | 50
  Between 18 and 65 years | 109 | 26485 | 26594
  >=65 years | 148 | 102072 | 102220
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (15.6) | 72.2 (11.5) | 72.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For the control group, the gender information was not available for all subjects in the CareLink database. Gender was unknown for 351 subjects in the control group.
  Participants
    number analyzed (Participants) | 257 | 128256 | 128513
    Female | 109 | 61604 | 61713
    Male | 148 | 66652 | 66800
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 152 | 128607 | 128759
  Italy | 12 | 0 | 12
  United Kingdom | 85 | 0 | 85
  France | 8 | 0 | 8
Education [Count of Participants; unit: Participants]
  Less Than High School | 17 | NA — This information is not available in CareLink database. | NA — Total not calculated because data are not available (NA) in one or more arms.
  High School | 111 | NA — This information is not available in CareLink database. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Bachelor | 86 | NA — This information is not available in CareLink database. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Master | 25 | NA — This information is not available in CareLink database. | NA — Total not calculated because data are not available (NA) in one or more arms.
  PhD/Doctorate | 18 | NA — This information is not available in CareLink database. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Chronic CareLink Transmission Success
Description: To assess CareLink transmission compliance (adherence to scheduled transmission), the primary objective is to compare the percentages of the CareLink quarterly scheduled transmissions that are completed within the prescribed window during the 12-month follow-up after the baseline visit in the CareLink Database between the evaluation patients who use the MyCareLink Heart™ (MCL) app and patients with low power devices and CareLink monitors 2490 (excluding wireless model 2490C). For both patient groups, all scheduled transmissions between 1 and 12 months after enrollment/CareLink activation were included.
  The results reflect the total percentage of completed transmissions pooled across subjects taking into account that there were several transmissions per subject. A correlated data method was required for the analysis. A 95% confidence interval based on generalized estimating equations for binomial distribution was calculated for the percentage of completed scheduled transmissions.
Time Frame: Scheduled transmissions between 1 and 12 months after enrollment/CareLink activation
Measure: Number (95% Confidence Interval); unit: Percentage of completed transmissions
Groups:
- Evaluation Group: Patients implanted with a pacemaker or CRT-P device who will be using remote monitoring via the MyCareLink Heart App
  Evaluation Group: Patient receiving exposure to the MyCareLink Heart App during device pairing
  Of the 257 enrolled patients, one patient was not available in CareLink database, 4 patients left evaluation early which resulted in data loss, 5 patients had no transmissions scheduled between 1 and 12 months, and 2 subjects had scheduled transmissions completed with another monitor than MyCareLink Heart App.
- Control Group (Historical): Patients with low power implantable devices and CareLink Monitor 2490 (Excluding wireless model 2490C)
  Control Group: Patients receiving exposure to the CareLink Monitor 2490 (Excluding wireless model 2490C)
  The enrolled patients in the evaluation were compared to a historical control group from the Medtronic de-identified CareLink™ database. The following inclusion criteria were used to select the analysis group from CareLink comparable to the BlueSync™ field evaluation : a) > 18 years of age at implant; b) Patient activated (first received CareLink transmission with CareLink 2490 monitor) in CareLink from 1 Jan 2016 to 1 December 2018; c) Patient followed for at least one year after activation with a minimum of one scheduled transmission in this year, d) US patients, e) Patient did not perform transmission with another monitor for at least one year after activation.
- Matched Control Group (Historical): Individual matching was performed using a greedy algorithm to create a matched control group comparable to the evaluation group. The matched control subjects were chosen from the historical control group with low power implantable devices and CareLink Monitor 2490 (excluding 2490C monitor).
  Subjects were matched exactly based on age (± 2 years), gender, and number of device chambers (single, dual or triple). For the evaluation group patients' age at screening was used while for the historical control cohort, age at implant was available. A range of two years was chosen since age at implant and age at screening should be within two years for the evaluation group with most patients having zero years between screening and implant.
Arm/Group | Evaluation Group | Control Group (Historical) | Matched Control Group (Historical)
Number analyzed (Participants) | 245 | 128607 | 979
Percentage of completed transmissions | 94.6 [91.8 to 96.6] | 60.0 [59.7 to 60.2] | 56.3 [53.7 to 58.9]
Statistical Analysis 1: Comparison: Evaluation Group vs Control Group (Historical); Test type: Superiority; p < 0.001, Generalized estimating equation model — The threshold for statistical significance was 0.025; Mean Difference (Final Values) = 34.7, 95% CI 2-sided [32.4 to 37.0]
Statistical Analysis 2: Comparison: Evaluation Group vs Matched Control Group (Historical); Test type: Superiority; p < 0.001, Generalized estimating equation model — The threshold for statistical significance was 0.025; Mean Difference (Final Values) = 38.3, 95% CI 2-sided [34.8 to 41.9]

2. Secondary Outcome: Acute CareLink Transmission Success
Description: To assess acute CareLink transmission compliance (adherence to scheduled transmission), the secondary objective is to characterize the percentage of the CareLink bi-weekly scheduled transmissions that are completed within the prescribed window during the 1-month follow-up after the baseline visit in the CareLink Database via the MCL Heart™ app. All scheduled transmissions within the first month after enrollment were included in the analysis.
  The results reflect the total percentage of completed transmissions pooled across all subjects taking into account that there were several transmissions per subject. A correlated data method was required for the analysis since there were several transmissions per subject. A two-sided 95% confidence interval based on generalized estimating equations (GEE) for binomial distribution was calculated for the percentage of completed scheduled transmissions.
Time Frame: Scheduled transmissions in the first month after enrollment
Population: In total, 215 patients had at least one scheduled transmission within the first month, and were available for analysis. Of the 257 enrolled patients, one patient was not available in CareLink, four patients left the evaluation early which resulted in data loss within CareLink, 37 patients had no scheduled transmission in the first month.
Measure: Number (95% Confidence Interval); unit: Percentage of completed transmissions
Arm/Group | Evaluation Group
Number analyzed (Participants) | 215
Percentage of completed transmissions | 95.1 [92 to 97]

ADVERSE EVENTS:
Time Frame: Not Collected
Description: Not Collected
Groups:
- Evaluation Group: Adverse events were not collected in the evaluation.
- Control Group (Historical): Adverse events are not available from the control group since the data of these patients is extracted from the Medtronic de-identified CareLink™ database.
Arm/Group | Evaluation Group | Control Group (Historical)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Version 1 (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT03518658/Prot_000.pdf
  • Study Protocol: Version 2 (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03518658/Prot_001.pdf
  • Study Protocol: Version 3 (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03518658/Prot_002.pdf
  • Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT03518658/SAP_003.pdf